CLINICAL TRIAL: NCT05688371
Title: Comparison of Addition of Dexmedetomidine to Low Dose Morphine Versus Standard Dose of Morphine in Patiant Controlled Analgesia in Children Undergoing Pelvi Abdominal Exploration. a Prospective Randomized Trial
Brief Title: Dexmedetomidine Plus Low Dose Morphine Versus Standard Dose of Morphine in PCA in Children .
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mariana Soliman, Benisuef university, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mariana AbdElsayed Mansour
Record Dates: First submitted 2022-12-25; First posted 2023-01-18 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-03

CONDITIONS: PCA; Children; Dexmedetomidine; Morphine
MeSH Terms: interventions — Morphine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard dose morphine (Active Comparator): children will receive 0.05 mg morphine /kg.as a bolus dose dissolved in 50 ml normal saline and 10 microgram/kg continuous infusion
  Interventions: Drug: standard dose morphine
- low dose morphine and dexmedetomidine (Active Comparator): children will receive 0.02 mg morphine /kg bolus dose plus 0.2 µg/kg dexmedetomidine dissolved in 50 ml normal saline and10 microgram/kg continuous infusion .
  Interventions: Drug: low dose morphine plus dexmedetomidine

INTERVENTIONS:
Drug: standard dose morphine — Receiving 0.05 mg morphine/kg as a bolus.
  Other Names: morphine sulphate
  Arms: standard dose morphine
Drug: low dose morphine plus dexmedetomidine — Receiving 0.02 mg morphine/kg as a bolus dose + 0.2 microgram/kg dexmedetomidine
  Other Names: precedex
  Arms: low dose morphine and dexmedetomidine

SUMMARY:
The treatment of perioperative pain in children has been a topic of great interest to pediatricians, pediatric surgeons, and anesthesiologists for many years. Opioids are the most common analgesics used to manage acute postoperative pain in children and adults

DETAILED DESCRIPTION:
Patient-controlled analgesia (PCA) permits patients to self-administer small doses of opioid analgesics intravenously or subcutaneously at frequent intervals. PCA is used in the management of moderate-to-severe pain. Patient-controlled analgesia (PCA) is now used in children as young as 5 yr for the treatment of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I & II of both sex.
2. Age between 8 and 12 years.
3. Patients scheduled for exploration surgery under general anesthesia.

Exclusion Criteria:

1. Parents refused to give consent.
2. Patients with history of allergy to morphine or dexmedetomidine.
3. Mental disorders.
4. Unsuitability for extubation.
5. Comorbidities as cardiac, pulmonary and obstructive sleep apnea.
6. children with chronic opioid use for > 3 monthes

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain intensity evaluation at (0,1, 2,6,12, 24h). | 24 hour
  visual analogue score consists of a straight 10 cm line with the end points defining extreme limits between (0) no pain and (10) worst pain, the score is determined by measuring the distance between no pain and worst pain.

SECONDARY OUTCOMES:
Total morphine consumption in 24h postoperative. | 24 hour
  total morphine dose in 24h
sedation | 24 hour
  (0 = awake; 1 = drowsy; 2 = asleep but arousable; 3 = deeply asleep). Patients were considered sedated if they had a sedation score of more than 0.
respiratory depression | 24 hour
  respiratory depression, if respiratory rate less than 10 breaths/minute
nausea vomiting | 24 hour
  Nausea and vomiting was recorded using a categorical scoring system (0 = none, 1 = nausea, 2 = retching, 3 = vomiting).

CONTACTS AND LOCATIONS:
Overall Officials: Mariana abdelsayed Mansour, Lecturer, Principal Investigator — Benisuef university hospital
Locations (1):
- Benisuef University Hospital, Egypt, Egypt